CLINICAL TRIAL: NCT06040112
Title: Effect of Atelocollagen Injection in Patients With Calcific Tendinitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hyungsuk Kim (Other)
Responsible Party: Sponsor-Investigator, Hyungsuk Kim, Assistant professor, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PC23DISV0050
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Calcific Tendinitis of Shoulder; Atelocollagen
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atelocollagen injection group (Experimental): Atelocollagen injection
  Interventions: Device: Atelocollagen
- Lidocain injection group (Placebo Comparator): Lidocain injection
  Interventions: Device: Atelocollagen

INTERVENTIONS:
Device: Atelocollagen — Tendoregen (Atelocollagen) injection
  Other Names: Tendoregen

SUMMARY:
Assess the clinical outcomes using atelocollagen injection in patients with calcific tendinitis.

DETAILED DESCRIPTION:
Suitable participants based on the selection/exclusion criteria are randomly assigned to either the case group or the control group. Consent is given right before the procedure.

Case group (Atelocollagen injection group): Ultrasound-guided barbotage followed by lidocaine and atelocollagen injection.

Control group (Lidocaine injection group): Ultrasound-guided barbotage followed by lidocaine injection."

Clinical outcomes will be assessed with functional scores on 6 months after injection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in whom calcification of 5mm or more is observed in plain radiographs.
2. In cases where concomitant medication is administered continuously during the clinical trial period, patients who have verified the exact prescribed medication taken within the last week and agreed to maintain the same amount throughout the study period.
3. Individuals who have agreed to participate in this study and have given written consent themselves.

Exclusion Criteria:

* Patients with a medical history of infectious arthritis, rheumatoid arthritis, tumors, or fractures.

  * Patients with hypersensitivity.

    * Patients with a history of anaphylactic reactions.

      * Patients with ongoing autoimmune diseases or a past medical history of such diseases, either in the patient or their family members.

        * Patients who are allergic to transplants. ⑥ Patients who are allergic to porcine (pig) proteins.

          ⑦ Patients deemed unsuitable for this trial based on the judgment of the trial administrator, such as those with mental illnesses.

          ⑧ Patients who have received intra-articular steroid or other injection treatments within one month prior to the procedure decision.

          ⑨ Patients who are on concomitant medications that include oral steroids.

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Constant score (Shoulder function score) | 1, 3, 5 months
  The Constant score is commonly used to evaluate the functional status of shoulder disorders and shows relatively high accuracy, reliability, and reproducibility. The evaluation is out of a total of 100 points: pain 15 points, daily activities 20 points, anterior elevation 10 points, lateral elevation 10 points, internal/external rotation each 10 points, and muscle strength 25 points

CONTACTS AND LOCATIONS:
Locations (1):
- Eunpyeong St. Mary's Hospital, The Catholic University of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No